CLINICAL TRIAL: NCT02760654
Title: Self-Guided Online Cognitive Behavioral Strategies for Chemotherapy-Induced Peripheral Neuropathy
Acronym: SONICS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: St. Joseph Mercy Health System (Unknown)
Responsible Party: Principal Investigator, Robert Knoerl, Dr., University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: HUM00104185
Record Dates: First submitted 2016-04-28; First posted 2016-05-03 (Estimated); Results first posted 2017-06-02 (Actual); Last update posted 2017-11-13 (Actual); Status verified 2017-10

CONDITIONS: Peripheral Nervous System Diseases; Pain Management; Self Management
MeSH Terms: conditions — Peripheral Nervous System Diseases; Agnosia

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Online Self Management (Experimental): Participants will interact with an online self management program based on cognitive behavioral principles for 8 weeks as much as they want.
  Interventions: Device: Proactive Self Management Program for Effects of Cancer Treatment
- Control (No Intervention): Treatment as usual

INTERVENTIONS:
Device: Proactive Self Management Program for Effects of Cancer Treatment
  Arms: Online Self Management

SUMMARY:
The purpose of this pilot randomized wait-list controlled trial is to test the efficacy of an online cognitive behavioral pain management website called Proactive Self-Management Program for Effects of Cancer Treatment (PROPSECT) to reduce worst pain intensity for individuals with chronic painful chemotherapy-induced peripheral neuropathy (CIPN) and to explore the mediating effect of PROSPECT-induced changes in anxiety, fatigue, depression, and sleep disturbance on worst pain intensity. Another aim of this study is to determine whether PROSPECT will decrease CIPN symptom severity (e.g. non-painful numbness and tingling), average pain severity, and physical impairment. Lastly, since this intervention has never been tested in individuals with painful CIPN, the investigators will assess patients' perceptions of acceptability and satisfaction with the intervention.

ELIGIBILITY:
Inclusion Criteria:

1. over 25 years of age
2. self-report 4/10 worst CIPN pain that has persisted three months or longer after the cessation of their neurotoxic chemotherapy regimen
3. have at least grade one sensory CIPN as defined by their oncology provider using the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE)
4. have a stable analgesic medication regimen as evidenced by a less than 10% increase or decrease in their analgesic medication dosage in the two weeks leading up to their enrollment in the study
5. have internet access
6. self-report the ability to use a computer
7. signed informed consent
8. willingness to participate in all study activities.

Exclusion Criteria:

1. prognosis of less than three months
2. documented peripheral neuropathy due to other causes (diabetes, alcohol abuse, Central Nervous System malignancy, vitamin B deficiency, hereditary, nerve compression injury)
3. neurotoxic chemotherapy treatment regimens are planned to occur while enrolled in the study
4. have participated in cognitive behavioral pain management in the past or plan to enroll in cognitive behavioral pain management during the course of the intervention.

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-04; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Knoerl, PhD, RN, Principal Investigator — University of Michigan
Locations (5):
- United States (5):
  - University of Michigan, Ann Arbor, Michigan
  - St. Joseph Mercy Canton, Canton, Michigan
  - St. Joseph Mercy Chelsea, Chelsea, Michigan
  - St. Joseph Mercy Livingston, Howell, Michigan
  - St. Joseph Mercy Ann Arbor, Ypsilanti, Michigan

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Online Self Management: Participants will interact with an online self management program based on cognitive behavioral principles for 8 weeks as much as they want.
  Proactive Self Management Program for Effects of Cancer Treatment
Period: Overall Study
Arm/Group | Online Self Management | Control
Started (Randomized) | 30 | 30
Completed | 23 | 24
Not Completed | 7 | 6
Not completed — Lost to Follow-up | 3 | 3
Not completed — Withdrawal by Subject | 4 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Online Self Management | Control | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.93 (9.33) | 63.37 (8.36) | 61.15 (9.06)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 22 | 45
  Male | 7 | 8 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 25 | 22 | 47
  Unknown or Not Reported | 5 | 7 | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 27 | 28 | 55
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 30 | 30 | 60
Education [Count of Participants; unit: Participants]
  High School or less | 4 | 6 | 10
  Some College | 13 | 12 | 25
  College Graduate | 8 | 6 | 14
  Post Graduate Degree | 5 | 5 | 10
  Missing/Unknown | 0 | 1 | 1
Employment Status [Count of Participants; unit: Participants]
  Employed | 13 | 7 | 20
  Out of Work | 3 | 2 | 5
  Homemaker | 0 | 1 | 1
  Retired | 9 | 17 | 26
  Unable to Work | 5 | 3 | 8
Marital Status [Count of Participants; unit: Participants]
  Single | 2 | 2 | 4
  Married | 18 | 24 | 42
  Separated | 1 | 1 | 2
  Divorced | 7 | 2 | 9
  Widowed | 2 | 1 | 3
Amount of Computer Use [Count of Participants; unit: Participants]
  Once a month | 1 | 6 | 7
  About once a week | 1 | 1 | 2
  More than once a week | 28 | 23 | 51
Cancer Stage [Count of Participants; unit: Participants]
  Early I-II | 13 | 9 | 22
  III | 10 | 11 | 21
  Metastatic (IV) | 6 | 9 | 15
  Unknown | 1 | 1 | 2
Cancer Type [Count of Participants; unit: Participants]
  Breast | 13 | 10 | 23
  Gastrointestinal | 13 | 13 | 26
  Lung | 1 | 3 | 4
  Multiple | 1 | 2 | 3
  Lymphoma | 2 | 1 | 3
  Genitourinary | 0 | 1 | 1
Chemotherapy Type [Count of Participants; unit: Participants]
  Platinums | 13 | 13 | 26
  Taxanes | 12 | 8 | 20
  Bortezomib | 1 | 0 | 1
  Vinca Alkaloids | 1 | 2 | 3
  Multiple | 3 | 7 | 10
Chemotherapy Name [Count of Participants; unit: Participants]
  Oxaliplatin | 13 | 13 | 26
  Paclitaxel | 9 | 4 | 13
  Docetaxel | 1 | 3 | 4
  Abraxane | 1 | 0 | 1
  Vincristine | 1 | 2 | 3
  Bortezomib | 1 | 0 | 1
  Multiple | 4 | 8 | 12
Pain-related Symptoms [Mean (Standard Deviation); unit: units on a scale] — Pain -related symptoms are measured from Patient Reported Outcome Measurement Information System surveys, and are measured along the following scales: Anxiety: 40.3 -81.6 where 40.3 means no anxiety to 81.6 as high anxiety. Depression: 41.0 -79.4 where 41 means no depression and 79.4 is ultimately high depression. Fatigue: 33.7 - 75.8 where 33.7 is no fatigue and 75.8 is extreme fatigue. Sleep related impairment: 30.0 - 80.1 where 30.0 is no impairment and 80.1 is high impairment in daily functioning due to poor sleep.
  units on a scale
    Anxiety (40.3 -81.6) | 54.79 (9.42) | 51.58 (7.83) | 53.18 (6.58)
    Depression (41.0 -79.4) | 52.92 (7.98) | 49.51 (7.17) | 51.22 (8.74)
    Fatigue (33.7 - 75.8) | 59.18 (8.26) | 52.73 (8.25) | 55.95 (7.71)
    Sleep-related Impairment (30.0 - 80.1) | 58.65 (6.67) | 55.07 (6.09) | 56.86 (8.81)

OUTCOME MEASURES:

1. Primary Outcome: Change in 0 - 10 Numerical Rating Scale of Worst Pain Intensity Scores at 8 Weeks
Description: Pain is measured on the numerical rating scale of 0 - 10 where 0 is no pain and 10 is worst imaginable pain.
Time Frame: Baseline to 8 weeks
Population: Only 19 people in each arm out of the 23 and 24 that completed the study actually completed the information for this measure. Thus only 19 are analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Online Self Management | Control
Number analyzed (Participants) | 19 | 19
units on a scale | -0.94 (1.36) | 0 (1.31)
Statistical Analysis 1: Comparison: Online Self Management vs Control; Test type: Superiority; p < 0.05, ANCOVA

2. Secondary Outcome: Change in PROMIS Short Form Emotional Distress - Depression 4a Scores at 8 Weeks
Description: The PROMIS short form emotional distress depression 4a Scores are measured on a scale whose lowest possible score is 41.0 and highest is 79.4 where 41 is no emotional distress and 79.4 is extreme distress.
Time Frame: Baseline to 8 weeks
Population: Only 19 in the people in the online self-management group and 23 in the Control group of the 23 and 24 that completed the study actually completed the information for this measure. Thus only 19 and 23 respectively are analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Online Self Management | Control
Number analyzed (Participants) | 19 | 23
units on a scale | -0.46 (6.15) | -1.27 (5.02)
Statistical Analysis 1: Comparison: Online Self Management vs Control; Test type: Superiority; p > 0.05, ANCOVA

3. Secondary Outcome: PROMIS Short Form Anxiety 4a
Description: The PROMIS Short Form Anxiety 4a is scored on a scale of 40.3 - 81.6, with a score of 40.3 meaning no anxiety and a score of 81.6 meaning high anxiety.
Time Frame: Baseline to 8 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Online Self Management | Control
Number analyzed (Participants) | 19 | 23
units on a scale | -1.26 (5.42) | -1.05 (8.46)
Statistical Analysis 1: Comparison: Online Self Management vs Control; Test type: Superiority; p > 0.05, ANCOVA

4. Secondary Outcome: Change in PROMIS Short Form Fatigue 4a Scores at 8 Weeks
Description: The PROMIS Short Form Fatigue 4a is scored on a scale of 33.7 to 75.8, with a score of 33.7 meaning no fatigue and a score of 75.8 meaning high fatigue.
Time Frame: Baseline to 8 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Online Self Management | Control
Number analyzed (Participants) | 19 | 23
units on a scale | -2.53 (5.99) | -1.69 (5.26)
Statistical Analysis 1: Comparison: Online Self Management vs Control; Test type: Superiority; p > 0.05, ANCOVA

5. Secondary Outcome: Change in PROMIS Short Form Sleep-Related Impairment 8a Scores at 8 Weeks
Description: The PROMIS Short Form Sleep-Related Impairment 8a is scored on a scale of 30.0 to 80.1 with a score of 30.0 meaning no sleep-related impairment and a score of 80.1 meaning a high degree of impairment in daily activities due to poor sleep.
Time Frame: Baseline to 8 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Online Self Management | Control
Number analyzed (Participants) | 19 | 23
units on a scale | -2.42 (4.05) | -1.29 (3.39)
Statistical Analysis 1: Comparison: Online Self Management vs Control; Test type: Superiority; p > 0.05, ANCOVA

6. Secondary Outcome: Patient Global Impression of Change
Description: The Patient Global Impression of Change is scored on a scale of 1 - 7, with a score of 1 representing that the patient was very much worse following the trial, and a score of 7 representing that the patient was very much improved following the course of the trial.
Time Frame: 8 week
Population: Only 19 in the people in the online self-management group and 22 in the Control group of the 23 and 24 that completed the study actually completed the information for this measure. Thus only 19 and 22 respectively are analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Online Self Management | Control
Number analyzed (Participants) | 19 | 22
Participants
  Improved | 9 | 6
  No Change/Worse | 10 | 16
Statistical Analysis 1: Comparison: Online Self Management vs Control; Test type: Superiority; p > 0.05, Fisher Exact

7. Secondary Outcome: Change in 0 - 10 Average Pain Intensity Numerical Rating Scale Scores at 8 Weeks
Description: The 0 - 10 Average Pain Intensity Numerical Rating Scale was scored on a scale of 0 - 10, with a score of 0 meaning no pain, and a score of 10 meaning worst pain imaginable.
Time Frame: Baseline to 8 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Online Self Management | Control
Number analyzed (Participants) | 19 | 23
units on a scale | 0.21 (2.59) | 1.44 (2.87)
Statistical Analysis 1: Comparison: Online Self Management vs Control; Test type: Superiority; p > 0.05, ANCOVA

8. Secondary Outcome: Adapted Acceptability E-Scale
Description: The Adapted Acceptability E- Scale contains 7 items that are scored on a 1 - 5 scale, with a score of 1 representing low ratings of acceptability and satisfaction with the online self management program, and a score of 5 representing high ratings of acceptability and satisfaction with the online self management program. This measure was only administered to individuals participating in the online self management program.
Time Frame: 8 week
Population: Only 19 in the people in the online self-management group of the 23 that completed the study actually completed the information for this measure. Thus only 19 are analyzed. No participants in the control group were administered this measure because the questions pertained to the acceptability and satisfaction of the online self management program.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Online Self Management | Control
Number analyzed (Participants) | 19 | 0
units on a scale
  How easy was it to access the website on your comp | 4.58 (0.84) |
  How understandable was the content presented withi | 4.58 (0.69) |
  How much did you enjoy using the website? | 3.26 (1.05) |
  How helpful was it to read and participate in the | 3.36 (0.96) |
  Was the amount of time it took to complete the act | 4 (1.11) |
  Was the amount of time it took to complete the stu | 4.42 (1.02) |
  Overall, how would you rate your satisfaction with | 3.95 (0.71) |
Statistical Analysis 1: Comparison: Online Self Management; Test type: Equivalence — Descriptive statistics (Mean, SD) were calculated for the 7 items of the Adapted Acceptability E-Scale; Calculated Mean and Standard Deviation = 0.05

9. Secondary Outcome: Change in European Organization of Research and Treatment of Cancer Quality of Life Questionnaire-Chemotherapy-Induced Peripheral Neuropathy Scale Scores at 8 Weeks
Description: The European Organization of Research and Treatment of Cancer Quality of Life Questionnaire-Chemotherapy-Induced Peripheral Neuropathy contains three subscales: Sensory, Motor, and Autonomic. Each subscale is scored on a scale of 0 - 100, with a score of 0 representing no neuropathy symptoms and functional impairment due to neuropathy, and a score of 100 represents severe neuropathy symptoms and functional impairment due to neuropathy. Only the Sensory and Motor subscales were used in this current study.
Time Frame: Baseline to 8 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Online Self Management | Control
Number analyzed (Participants) | 19 | 23
units on a scale
  Sensory Subscale | -8.93 (17.69) | 4.04 (13.57)
  Motor Subscale | -7.3 (15.6) | -3.08 (14.37)
Statistical Analysis 1: Comparison: Online Self Management vs Control; Test type: Superiority; p > 0.05, ANCOVA

10. Secondary Outcome: Change in PROMIS Pain Interference 4a Scores at 8 Weeks
Description: The PROMIS Pain Interference 4a is scored on a scale of 41.6 to 75.6, with a score of 41.6 meaning little or no interference with daily activities due to pain severity, and a score of 75.6 meaning a high degree of interference with daily activities due to pain severity.
Time Frame: Baseline to 8 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Online Self Management | Control
Number analyzed (Participants) | 19 | 23
units on a scale | -1.10 (7.58) | -0.89 (2.89)
Statistical Analysis 1: Comparison: Online Self Management vs Control; Test type: Superiority; p > 0.05, ANCOVA

ADVERSE EVENTS:
Time Frame: Adverse event data was collected from the Baseline (Time of randomization) to the Week 8 (Final) time points.
Description: We called participants 4 and 8 weeks after beginning the study to ask them if they experienced any negative effects from participating in the study.
Arm/Group | Online Self Management | Control
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30

LIMITATIONS AND CAVEATS:
Small sample size, high drop out, lack of active monitoring of intervention usage, lack of generalizability to any specific type of chronic painful neuropathy, and changes in pain medications during the trial may have confounded the primary analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No